CLINICAL TRIAL: NCT02792569
Title: Auto-transplantation of Fragmented Ovarian Cortical Tissue in Infertile Patients With Premature Ovarian Oocyte Depletion - a Study to Promote Follicular Activation and Subsequent Fertility
Brief Title: Follicle Activation by Inhibition of the Hippo Pathway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anders Nyboe Andersen (Other)
Responsible Party: Sponsor-Investigator, Anders Nyboe Andersen, Professor M.D., Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-15011975
Record Dates: First submitted 2016-05-23; First posted 2016-06-07 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Infertility
Keywords: IVA; Hippo Pathway; Follicle activation; Low Responder; POI; Poor Ovarian Reserve; Poor Ovarian Response; Salvador/Warts/Hippo pathway
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biopsy at Right side (Experimental): Biopsy of ovarian cortical tissue (50% right side)
  Interventions: Procedure: Biopsy of ovarian cortical tissue
- Biopsy at Left side (Experimental): Biopsy of ovarian cortical tissue (50% left side)
  Interventions: Procedure: Biopsy of ovarian cortical tissue

INTERVENTIONS:
Procedure: Biopsy of ovarian cortical tissue — Biopsies will be taken from either right or left side. The cortical tissue will be isolated and fragmented in 1x1 mm2 pieces, followed by auto-transplantation to a peritoneal pocket.

SUMMARY:
The aim of this project is to activate recruitment and growth of resting primordial follicles in the ovaries of women with diminished ovarian reserve, in attempt to increase the chance to become pregnant, either naturally or after assisted reproduction.

DETAILED DESCRIPTION:
For this study investigators will carefully select 20 women with low AMH and imminent POI.

They will be randomized to have cortical ovarian biopsies taken from either the left or right ovary. The biopsies will be fragmented in 1x1 mm2 pieces and immediately auto-transplanted in a peritoneal pocket under the right ovary.

The contralateral untouched ovary will act as the control, making each woman their own control.

Follow up: each week in 2,5 months the women will be assessed by transvaginal ultrasound and hormonal status. After 2,5-6 months the women will receive a FSH stimulation cycle (rFSH 300 IU or Corifollitropin) followed by standard IVF/ICSI,

Hypothesis: the ovaries contain a pool of resting primordial follicles. By fragmentation of cortical ovarian tissue, manipulation of the local environment in the tissue will inhibit the Hippo Pathway and hereby active recruitment and growth of primordial follicles.

ELIGIBILITY:
Inclusion Criteria:

* Infertility with indication for IVF/ICSI
* Imminent POI, still cycling
* Age 25 - 39 years
* Two ovaries
* Serum AMH measurements < 5 pmol/l (two independent measurements)
* Antral follicle count (AFC) (sum of both ovaries < 5)

Exclusion Criteria:

* Ovarian pathology (endometriosis, cysts)
* Known chromosomal abnormality
* Known autoimmune disease (except TPO-antibodies)
* Patients who have contraindication for laparoscopy

Ages: 25 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-04; Primary Completion 2018-12 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Number of follicles > 12 mm | Up to 6 month after the auto-transplantation
  Number of follicles > 12 mm in response to controlled ovarian stimulation with corifollitropin from the biopsied ovary versus the contralateral untreated ovary

SECONDARY OUTCOMES:
Side of ovulation | Up to 6 months after auto-transplantation
  Frequency of ovulations occurring at the "biopsy side" versus the contralateral side in the subsequent 4- 6 months

OTHER OUTCOMES:
AFC count | Up to 10 month after auto-transplantation
  Number of antral follicles (AFC) at the biopsy side versus that of the contralateral side
AMH changes | Up up to 10 month after auto-transplantation
  Changes (increase - decrease) in serum AMH over time, using the highly sensitive new AMH Assay (Elecsys Assay; Roche), which has been implemented as a routine analysis at The Department of Clinical Biochemistry Rigshospitalet in June 1st 2015
Pregnancy | Through study completion, an average of 1 year
  Numbers of pregnancies (spontaneously/assisted)

CONTACTS AND LOCATIONS:
Overall Officials: Anders N Andersen, Professor, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- The Fertility Clinic, Rigshospitalet, Copenhagen University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kawamura K, Cheng Y, Suzuki N, Deguchi M, Sato Y, Takae S, Ho CH, Kawamura N, Tamura M, Hashimoto S, Sugishita Y, Morimoto Y, Hosoi Y, Yoshioka N, Ishizuka B, Hsueh AJ. Hippo signaling disruption and Akt stimulation of ovarian follicles for infertility treatment. Proc Natl Acad Sci U S A. 2013 Oct 22;110(43):17474-9. doi: 10.1073/pnas.1312830110. Epub 2013 Sep 30. PMID 24082083
- [Background] Hsueh AJ, Kawamura K, Cheng Y, Fauser BC. Intraovarian control of early folliculogenesis. Endocr Rev. 2015 Feb;36(1):1-24. doi: 10.1210/er.2014-1020. Epub 2014 Sep 9. PMID 25202833
- [Background] Suzuki N, Yoshioka N, Takae S, Sugishita Y, Tamura M, Hashimoto S, Morimoto Y, Kawamura K. Successful fertility preservation following ovarian tissue vitrification in patients with primary ovarian insufficiency. Hum Reprod. 2015 Mar;30(3):608-15. doi: 10.1093/humrep/deu353. Epub 2015 Jan 6. PMID 25567618
- [Derived] Lunding SA, Pors SE, Kristensen SG, Landersoe SK, Jeppesen JV, Flachs EM, Pinborg A, Macklon KT, Pedersen AT, Andersen CY, Andersen AN. Biopsying, fragmentation and autotransplantation of fresh ovarian cortical tissue in infertile women with diminished ovarian reserve. Hum Reprod. 2019 Oct 2;34(10):1924-1936. doi: 10.1093/humrep/dez152. PMID 31593582